CLINICAL TRIAL: NCT01041937
Title: Total Knee Arthroplasty Randomized Clinical Trial- Cemented vs. Cementless Tibial Prosthesis Study
Brief Title: Total Knee Arthroplasty (TKA) Cemented Versus Cementless Tibial Prosthesis Study
Acronym: TKA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Stryker Trauma and Extremities (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Clohisy TKA trial-201102554
Record Dates: First submitted 2010-01-04; First posted 2010-01-05 (Estimated); Last update posted 2019-01-08 (Actual); Status verified 2019-01

CONDITIONS: Osteoarthritis; Post-traumatic Osteoarthritis; Rheumatoid Arthritis
MeSH Terms: conditions — Osteoarthritis; Arthritis, Rheumatoid

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cemented Tibia (Active Comparator): Assessing the clinical outcomes of the different type of fixation
  Interventions: Procedure: Cemented Tibia
- Cementless Tibia (Active Comparator): Assessing the clinical outcomes of the different type of fixation
  Interventions: Procedure: Cementless Tibia

INTERVENTIONS:
Procedure: Cemented Tibia — Total knee arthroplasty with cemented or cemented tibia, and post operative clinical outcome tracking
  Arms: Cemented Tibia
Procedure: Cementless Tibia — Assessing the clinical outcomes of the different type of fixation
  Arms: Cementless Tibia

SUMMARY:
The primary purpose of TKA Randomized Clinical Trial- Cemented versus Cementless Tibial Prosthesis Study will determine whether there is a significant difference in patient-reported and measured clinical outcomes (e.g. pain, function, length of recovery, and patient satisfaction) between subjects treated with a cementless tibial prosthesis (the cementless group) and those treated with cemented tibial prosthesis (the cement group) over the first two postoperative years. Radiographs will be assessed before surgery and at established post-operative intervals to determine if there are any significant differences between patients in the two groups and to assess the influence of component fixation on radiographic stability over time. Complication and revision rates will also be assessed for comparison.

ELIGIBILITY:
Inclusion Criteria:

* BMI less than <35
* Normal neurological function
* Primary total knee arthroplasty (Pre operative Medial Knee Patient)
* Patient age ≤ 70 years old

Exclusion Criteria:

* Revision surgery
* History of joint sepsis
* Recent systemic corticosteroids (< 2 months prior to procedure)
* Primary or secondary carcinoma in the last five years
* Post operative renal transplant
* Psychosocial disorders limiting rehabilitation
* Previous intraarticular knee fracture
* Over 20° valgus or varus deformity
* Extension loss over 20°
* Unsuitable for cruciate- substituting arthroplasty
* Unsuitable for cementless fixation of the tibial component
* Need for augmentation wedges or bone graft
* Previous proximal tibial osteotomy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2009-12; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
To use clinical outcome measures to assess for differences in patient function, quality of life and satisfaction between patients who have tibial component placement with either a cemented or a cementless technique | 2014

CONTACTS AND LOCATIONS:
Overall Officials: John Clohisy, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States